CLINICAL TRIAL: NCT03845153
Title: Study of Metformin Drug Effect on Fracture Healing in Post-Menopausal Women and Its Correlation to Serum Irisin Myokine Level.
Brief Title: Metformin Effect on Fracture Healing in Post-Menopausal Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Damanhour University (Other)
Responsible Party: Principal Investigator, Rehab Werida, Principal Investigator, Damanhour University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Metformin on Fracture healing
Record Dates: First submitted 2019-02-15; First posted 2019-02-19 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Bone Fracture
Keywords: Bone Fracture; Post-Menopausal Women; Metformin; Irisin
MeSH Terms: conditions — Fractures, Bone | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: 40 post-menopausal women with a bone fracture divided into two groups each of 20, randomly assigned to administration with metformin Retard 850 mg once daily for two weeks then 850 mg twice daily or with placebo.
Who Masked: Participant, Outcomes Assessor
Masking Description: double-blind perspective study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin (Active Comparator): 20 post-menopausal women with a bone fracture treated with metformin Retard 850 mg once daily for two weeks then 850 mg twice daily for three months.
  Interventions: Drug: Metformin Retard 850 mg
- Placebo (Placebo Comparator): 20 post-menopausal women with a bone fracture treated with placebo once daily for two weeks then twice daily for three months.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Metformin Retard 850 mg — tablet
  Other Names: Glucophage
  Arms: Metformin
Other: Placebo — placebo tablet
  Arms: Placebo

SUMMARY:
study the effect of metformin drug on fracture healing of patients with high risk of delayed fracture healing or non-union and correlating this to serum irisin myokine level.

DETAILED DESCRIPTION:
1. Approval will be obtained from Ethics Committee of general organization of teaching hospitals and institutes and Research Ethics Committee of Faculty of Pharmacy, Damanhour University.
2. Getting informed consent from all participants to take part in this study.
3. Two groups each of 20 post-menopausal women with a bone fracture. One group will be treated randomly with metformin Retard 850 mg once daily for two weeks then 850 mg twice daily. The other group will be untreated and served as control group.
4. Venous blood samples will be taken from each patient before fracture stabilization and later for determination of serum irisin level with corresponding radiological evaluations.

Inclusion criteria:

• Age range from 55 to less than 65 years old with bone fracture.

Exclusion criteria:

* Age equal or less than 55 years
* Age equal or more than 65 years
* Unstable or hospitalized patients with heart failure
* Hepatic impairment
* Chronic kidney disease with eGFR <45 mL/minute/1.73 m2
* Open fractures
* Pathological fractures
* Diabetic patients Statistical tests appropriate to the study design will be conducted to evaluate the significance of the results.

Methodology:

* Active Human Irisin ELISA kit will be used.
* Bone-specific Alkaline phosphatase BAP
* Serum creatinine, serum albumin, prothrombin time.
* Fasting insulin, fasting blood glucose and Calcium level.
* BMI, weight, waist, waist-hip ratio, total cholesterol and low-density-lipoprotein cholesterol.
* radiological scoring system will be used to evaluate the degree of new bone formation in the fracture line on anterior-posterior and lateral radiographs will be taken two months post stabilization.

ELIGIBILITY:
Inclusion Criteria:

* Age range from 55 to less than 65 years old with bone fracture.

Exclusion Criteria:

* Age equal or less than 55 years
* Age equal or more than 65 years
* Unstable or hospitalized patients with heart failure
* Hepatic impairment
* Chronic kidney disease with eGFR <45 mL/minute/1.73 m2
* Open fractures
* Pathological fractures
* Diabetic patients

Ages: 55 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — post-menopausal women
Enrollment: 40 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Human Irisin (ng/ml) | three months
  myokine/adipokine
Bone specific alkaline phosphatase (IU/L) | three months
  isoenzyme produced by osteoblasts involved with calcification of skeleton and bone formation
postoperative X-rays - Lane and Sandhu radiological scoring system | two months post stabilization.
  evaluate the degree of new bone formation in the fracture line on anterior-posterior and lateral radiographs

CONTACTS AND LOCATIONS:
Overall Officials: Gamal Omran, Professor, Study Director — Damanhour University
Locations (1):
- Damanhour Medical National Institute, Damanhūr, El-Bahairah, Egypt

IPD SHARING:
Plan to Share IPD: No